CLINICAL TRIAL: NCT02573948
Title: Feasibility of an Interventional Project to Reduce HIV Incidence Among People Who Inject Drugs in Haiphong, Viet Nam
Brief Title: Feasibility of Interventions on People Who Inject Drugs in Vietnam
Acronym: DRIVE-IN
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANRS12299 DRIVE IN; P30DA011041 (NIH)
Record Dates: First submitted 2015-09-22; First posted 2015-10-12 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: HIV; Hepatitis Virus; Substance Abuse
Keywords: People who inject drugs; Vietnam; Community support groups
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention is assessed

SUMMARY:
This study aims at assessing the feasibility of implementing an interventional cohort of people who inject drugs in Haiphong, Viet Nam.

For this purpose, the investigators will conduct a RDS survey to i) assess the current situation of drug use behaviour, HIV and Hepatitis C Virus (HCV) infection in the study population and ii) recruit participants for the longitudinal phase. The latter will consist of enroling the most difficult to reach People Who Inject Drugs (PWID) (those not followed by health centers), including early injectors, Men who have Sex with Men (MSM) and female sex workers (FSW) and following them up for 6 months in order to estimate the follow-up rate and preliminary estimates of HIV and HCV incidence.

DETAILED DESCRIPTION:
Objectives:

The primary objective of the DRIVE-IN project is to evaluate the feasibility of implementing an interventional cohort of PWID in Haiphong. Such a cohort (DRIVE) will be instrumental in demonstrating the efficacy of a community-involved intervention integrating prevention and care in order to reduce HIV and HCV transmission among PWID in Haiphong.

The main expected result of DRIVE-IN is to demonstrate that enrolment and follow-up of various hard-to-reach subgroups of PWID is feasible in the local context. These feasibility objectives will be evaluated using a set of relevant indicators.

Design:

The research will first include a respondent-driven sampling (RDS) survey, including a maximum of 600 PWID. Then 250 RDS participants (i.e about a quarter of the future DRIVE cohort) will be selected for a longitudinal study, with an enrolment and 3 follow-up visits at week 4, 12 and 24. In parallel, four qualitative studies will be implemented: one study to explore how to reach the hardest-to-reach and most-at-risk PWID, one feed-back study on PWID feeling about their participation in the research, one study investigating the reasons of drop-outs, and a final study on the research process itself.

Endpoints:

The RDS will describe the target population and the patterns of drug use. The feasibility of implementing an interventional cohort will be evaluated on several indicators:

* International multi-disciplinary research network is operational
* Completion of recruitment within the time frame
* Follow-up rate >80% at 24 weeks
* Implementation and increased access to peer-led interventions
* Establishment of a data management center
* Improved laboratory capacities for research
* Documented support of local and national authorities

Study population RDS survey Inclusion criteria Age > 18 years Self-reported drug injector confirmed by a positive urinary test and either skin marks of injection or knowledge of injecting procedures Signed informed consent Non-inclusion criteria Unable of understanding informed consent and answering questionnaires

Longitudinal study Inclusion criteria Having participated to the RDS survey Signed informed consent specific to the longitudinal study Non-inclusion criteria Ongoing Methadone Maintenance Therapy (MMT) Ongoing antiretroviral therapy Health status not compatible with study follow-up Have a plan to move out of Haiphong over the next two years. Have been sentenced recently to a prison term

Follow-up and study visits contents:

Participants of the longitudinal phase will be followed at week 4, 12 and 24 (final visit). During the RDS, face-to-face questionnaires will be applied on drug use, sexual health, and referral to care and repeated at each follow-up visit, along with the record of medical events. In addition, a urinary test will be collected at the RDS to assess the range of recent drugs used, and repeated at the final follow-up visit (week 24). Finally, at the RDS and final visit, HIV, HCV, Hepatitis B Virus (HBV) serology will be done along with appropriate counselling.

Sample size:

* 603 PWID will be enrolled in the RDS survey
* 250 RDS participants will be enroled in the longitudinal phase, including:
* 140 PWID for > 2 years, including females
* 50 recent injectors (< 2 years from first injection)
* 30 FSW who inject drugs
* 30 MSM who inject drugs

ELIGIBILITY:
* Inclusion criteria

  * Being more than 18 years of age
  * Being drug injector confirmed by a positive urine drug test with knowledge of injecting procedures
  * Having signed the informed consent form
  * For the Longitudinal study - having participated in the RDS survey
* Exclusion criteria

  * Unable to understand informed consent and how to answer a questionnaire
  * For the longitudinal study - being under methadone maintenance therapy and antiretroviral treatment
  * Having a health condition not compatible with study follow-up
  * Plan to move away from Haiphong in the next 2 years
  * Serving a sentence in prison

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who inject drugs living in Haiphong, Vietnam. The longitudinal phase will be restricted to those not followed by health care services, i.e. not taking methadone nor antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Nagot, MD,PhD, Principal Investigator — INSERM U1058 & University of Montpellier, France; Oanh Khuat Thi, MD, MSc, Principal Investigator — Supporting Community Development Initiatives (SCDI); Don DesJarlais, PhD, Principal Investigator — Mount Sinai Beth Israel
Locations (1):
- Hai Phong Medical University, Haiphong, Vietnam

REFERENCES:
- [Background] Elliott JC, Hasin DS, Stohl M, Des Jarlais DC. HIV, Hepatitis C, and Abstinence from Alcohol Among Injection and Non-injection Drug Users. AIDS Behav. 2016 Mar;20(3):548-54. doi: 10.1007/s10461-015-1113-z. PMID 26080690
- [Background] Perlman DC, Des Jarlais DC, Feelemyer J. Can HIV and Hepatitis C Virus Infection be Eliminated Among Persons Who Inject Drugs? J Addict Dis. 2015;34(2-3):198-205. doi: 10.1080/10550887.2015.1059111. PMID 26075647
- [Background] Perlman DC, Jordan AE, Uuskula A, Huong DT, Masson CL, Schackman BR, Des Jarlais DC. An international perspective on using opioid substitution treatment to improve hepatitis C prevention and care for people who inject drugs: Structural barriers and public health potential. Int J Drug Policy. 2015 Nov;26(11):1056-63. doi: 10.1016/j.drugpo.2015.04.015. Epub 2015 Apr 27. PMID 26050614
- [Background] Hatzakis A, Sypsa V, Paraskevis D, Nikolopoulos G, Tsiara C, Micha K, Panopoulos A, Malliori M, Psichogiou M, Pharris A, Wiessing L, van de Laar M, Donoghoe M, Heckathorn DD, Friedman SR, Des Jarlais DC. Design and baseline findings of a large-scale rapid response to an HIV outbreak in people who inject drugs in Athens, Greece: the ARISTOTLE programme. Addiction. 2015 Sep;110(9):1453-67. doi: 10.1111/add.12999. Epub 2015 Jul 14. PMID 26032121
- [Background] Des Jarlais DC. AIDS, people who use drugs, and altruism: reflection on a personal image. Subst Use Misuse. 2015 Mar;50(4):532-3. doi: 10.3109/10826084.2015.978185. Epub 2014 Dec 26. No abstract available. PMID 25540950
- [Result] Michel L, Des Jarlais DC, Duong Thi H, Khuat Thi Hai O, Pham Minh K, Peries M, Vallo R, Nham Thi Tuyet T, Hoang Thi G, Le Sao M, Feelemyer J, Vu Hai V, Moles JP, Laureillard D, Nagot N; DRIVE Study Team. Intravenous heroin use in Haiphong, Vietnam: Need for comprehensive care including methamphetamine use-related interventions. Drug Alcohol Depend. 2017 Oct 1;179:198-204. doi: 10.1016/j.drugalcdep.2017.07.004. Epub 2017 Aug 2. PMID 28800503
- [Result] Des Jarlais D, Duong HT, Pham Minh K, Khuat OH, Nham TT, Arasteh K, Feelemyer J, Heckathorn DD, Peries M, Moles JP, Laureillard D, Nagot N; (The Drive Study Team). Integrated respondent-driven sampling and peer support for persons who inject drugs in Haiphong, Vietnam: a case study with implications for interventions. AIDS Care. 2016 Oct;28(10):1312-5. doi: 10.1080/09540121.2016.1178698. Epub 2016 May 13. PMID 27178119
- [Result] Des Jarlais DC, Thi Huong D, Thi Hai Oanh K, Khue Pham M, Thi Giang H, Thi Tuyet Thanh N, Arasteh K, Feelemyer J, Hammett T, Peries M, Michel L, Vu Hai V, Roustide MJ, Moles JP, Laureillard D, Nagot N; DRIVE Study Team. Prospects for ending the HIV epidemic among persons who inject drugs in Haiphong, Vietnam. Int J Drug Policy. 2016 Jun;32:50-6. doi: 10.1016/j.drugpo.2016.02.021. Epub 2016 Feb 27. PMID 27006257
- [Result] Duong HT, Jarlais DD, Khuat OHT, Arasteh K, Feelemyer J, Khue PM, Giang HT, Laureillard D, Hai VV, Vallo R, Michel L, Moles JP, Nagot N; Drive Study Group. Risk Behaviors for HIV and HCV Infection Among People Who Inject Drugs in Hai Phong, Viet Nam, 2014. AIDS Behav. 2018 Jul;22(7):2161-2171. doi: 10.1007/s10461-017-1814-6. PMID 28612212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: People Who Injected Drugs (PWID), age > 18 years, with history of injecting drug use confirmed by a positive urine test and visual inspection of injection marks
Groups:
- People Who Injected Drugs (PWID) Respondent Driven Sample (RDS: 603 participants recruited through Respondent Driven Sample survey
Period: RDS
Arm/Group | People Who Injected Drugs (PWID) Respondent Driven Sample (RDS
Started | 603
Completed | 603
Not Completed | 0
Period: Longitudinal Cohort
Arm/Group | People Who Injected Drugs (PWID) Respondent Driven Sample (RDS
Started (Among 603 RDS participants, 250 PWID were selected for the longitudinal follow-up.) | 250 (Not on ART a/o MMT. MSM and FSW were prioritized for enrolling,)
Completed | 194
Not Completed | 56
Not completed — Death | 9
Not completed — Lost to Follow-up | 22
Not completed — Incarcerated | 25

BASELINE CHARACTERISTICS:
Groups:
- PWID RDS: 603 participants
Arm/Group | PWID RDS
Number analyzed (Participants) | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 542
Region of Enrollment [Number; unit: participants]
  Vietnam | 603
Medical Insurance [Count of Participants; unit: Participants] | 105
Duration of Injection use [Median (Inter-Quartile Range); unit: years] | 8 [4 to 13]
Number of drug injection (typical day) [Mean (Standard Deviation); unit: injection per day] | 2.7 (1)
Injecting drug: heroin alone [Count of Participants; unit: Participants] | 602
Injection with syringe already used by someone else (last 3 months) [Count of Participants; unit: Participants] | 33
HIV positive [Count of Participants; unit: Participants] | 152
Currently under Methadone Maintenance Therapy [Count of Participants; unit: Participants] | 36
HCV positive [Count of Participants; unit: Participants] | 398

OUTCOME MEASURES:

1. Primary Outcome: Number of Cohort Participants Attending the Last Follow-up Visit at W52
Description: Number of participants who were followed up and not lost to follow-up after enrolment into cohort.
Time Frame: 52 weeks
Population: Participants were invited to follow-up visits at W4, W12, W24 and W52
Measure: Count of Participants; unit: Participants
Groups:
- PWID Cohort: 250 participants selected among 603 RDS participants
Arm/Group | PWID Cohort
Number analyzed (Participants) | 250
Participants | 194

2. Secondary Outcome: HCV Seroconversion
Description: Number of new HCV infection among HCV negative (at RDS) cohort participants over 1 year period
Time Frame: 52 weeks
Population: HCV negative cohort participants with HCV test result available at W24 and/or W52.
Measure: Count of Participants; unit: Participants
Groups:
- HCV Negative Cohort Participants: Cohort participants, HCV negative at RDS
Arm/Group | HCV Negative Cohort Participants
Number analyzed (Participants) | 92
Participants | 18

3. Secondary Outcome: HIV Seroconversion
Description: Number of new HIV infection among HIV negative (at RDS) cohort participants over 1 year period.
Time Frame: 52 weeks
Population: HIV negative cohort participants with HIV test result available at W24 and/or W52.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Negative Cohort Participants: Cohort participants, HIV negative at RDS.
Arm/Group | HIV Negative Cohort Participants
Number analyzed (Participants) | 180
Participants | 0

4. Secondary Outcome: Incidence of HCV Infection
Description: The HCV incidence was calculated by 100person/year
Time Frame: 52 weeks
Population: HCV negative cohort participants with HCV test result available at W24 a/or W52
Measure: Number (95% Confidence Interval); unit: infections per 100 person-years
Groups:
- HCV Negative Cohort Participants: HCV negative (at RDS) participants
Arm/Group | HCV Negative Cohort Participants
Number analyzed (Participants) | 92
infections per 100 person-years | 19.4 [11.5 to 30.7]

5. Secondary Outcome: HIV Incidence
Description: HIV incidence was calculated by 100person/year. With zero conversion, we choose 2.5% unilateral confidence interval.
Time Frame: 52 weeks
Population: HIV negative cohort participants with HCV test result available at W24 a/or W52
Measure: Number (2.5% Confidence Interval); unit: infections per 100 person-years
Arm/Group | HIV Negative Cohort Participants
Number analyzed (Participants) | 180
infections per 100 person-years | 0 [0 to 1.8]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Adverse events reported for cohort participants (n=250)
Groups:
- PWID Cohort: 250 participants
Arm/Group | PWID Cohort
All-Cause Mortality (participants affected / at risk) | 9/250
Serious Adverse Events (participants affected / at risk) | 9/250
Other Adverse Events (participants affected / at risk) | 0/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PWID Cohort (N=250)
Overdose (General disorders) | 2 (2)
AIDS (Immune system disorders) | 5 (5)
Suicide (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No